CLINICAL TRIAL: NCT05862584
Title: Impact of Air Pollution on the Course of Inflammatory Rheumatism: a Prospective, Single-center Study
Brief Title: Impact of Air Pollution on the Course of Inflammatory Rheumatism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-PP-02
Record Dates: First submitted 2023-04-24; First posted 2023-05-17 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-03

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main Cohort (Experimental): Cohort of patients with inflammatory rheumatism (rheumatoid arthritis or spondyloarthritis diagnosed according to ACR/EULAR 2010 or ASAS), over 18 years of age, and with stable chronic inflammatory rheumatism under biological treatment
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Distribution of questionnaires to patients to be completed on a weekly basis.

SUMMARY:
The objective of this study is to see if there is a link between air pollution and inflammatory rheumatism (rheumatoid arthritis and ankylosing spondylitis)

To do this, the investigators are going to follow a cohort of about 200-400 patients for 6 months by means of a self-questionnaire, which the investigators ask the patient to fill in once a week on a fixed day, and opposite the corresponding week to put the letter corresponding to the question concerning the activity of your disease: 3 possible answers: A: no flare-up, B: short flare-up of 1 to 3 days, C: persistent flare-up of more than 3 days

Then the investigators will collect the questionnaire at the end of these 6 months and at each visit to the consultation or day hospital (on average every 4 to 6 weeks), and they will look to see if any relapses have occurred. At the same time the investigators will calculate the disease activity score (DAS or BASDAI) to have an objective score. Then in parallel they will look at the level of exposure to air pollution according to the place of residence and work of each patient.

The hypothesis is that air pollution has an influence on the activity of inflammatory rheumatism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA according to ACR/EULAR 2010 criteria, or spondyloarthritis according to ASAS criteria.
* Patients older than 18 years of age
* Patients with RA or spondyloarthritis considered stable (no change in background or biological therapy for at least 3 months) and in low activity (SAR 28 CRP < 3.2 for RA and BASDAI < 4 for 3 months).
* Patient treated with biological therapy

Exclusion Criteria:

* Patient with no fixed abode
* Patient planning to move within 6 months.
* Patient unable to read or understand the non-opposition notice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Show that there is a difference in average exposure to regulated pollutants according to the occurrence or non-occurrence of inflammatory rheumatism (RA or APS). | Every week for 6 months
  Occurrence of a flare-up of less than 3 days and/or more than 3 days

SECONDARY OUTCOMES:
Relationship between average exposure to regulated pollutants and severity of SPA/PR. | Every week for 6 months
  The relationship between average exposure to regulated pollutants and severity (duration of flare) of SPA/PR data of flare-up of less than 3 days and/or more than 3 days will be collected with questionnaires.
Correlations between average exposure to regulated pollutants and biological severity of SPA/PR. | Every week for 6 months
  Correlations between average exposure to regulated polluants and biological severity data of flare-up of less than 3 days and/or more than 3 days will be collected with questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No